CLINICAL TRIAL: NCT02318069
Title: Humoral Response to TBE Vaccine in Elderly (50+ Year Olds) After Changed Dosage Intervals/Number of Doses?
Brief Title: New Study - Humoral Response to Tick-borne Encephalitis Vaccine in Elderly
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Sormland County Council, Sweden (Other)
Collaborators: Karolinska Institutet (Other); Helsingfors university (Unknown)
Responsible Party: Principal Investigator, Lars Rombo, professor, Sormland County Council, Sweden
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2011/4-31/2 - B
Record Dates: First submitted 2014-12-12; First posted 2014-12-17 (Estimated); Last update posted 2021-02-10 (Actual); Status verified 2021-02

CONDITIONS: Tick-borne Encephalitis
Keywords: immune response; TBE-vaccine; elderly; additional doses
MeSH Terms: conditions — Encephalitis, Tick-Borne

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- TBE vaccine at 0+30 days (Active Comparator): This group of 50 participants will follow the standard recommendation and will be given TBE vaccine 0.5 ml FSME immune at 0 + 30 days during the first year and an additional dose one year later
  Interventions: Biological: FSME-immune
- TBE vaccine at 0+7+21 days (Active Comparator): This group of 50 participants will will be given TBE vaccine 0.5 ml FSME immune at 0 + 7 +21 days during the first year and an additional dose one year later
  Interventions: Biological: FSME-immune
- TBE vaccine at 0+30+90 days (Active Comparator): This group of 50 participants will will be given TBE vaccine 0.5 ml FSME immune at 0 + 30 + 90 days during the first year and an additional dose one year later
  Interventions: Biological: FSME-immune
- younger participants (Active Comparator): This group of 50 participants in the age group 18-49 years will be given TBE vaccine 0.5 ml FSME immune at 0 +30 days during the first year and an additional dose one year later
  Interventions: Biological: FSME-immune
- double dose of vaccine (Active Comparator): This group of 50 participants will be given two doses of TBE vaccine 0.5 ml FSME immune at the first day of the study and an additional dose at day 30 as well as one year later
  Interventions: Biological: FSME-immune

INTERVENTIONS:
Biological: FSME-immune — 0.5 ml im as scheduled in the 5 arms

SUMMARY:
The risk for tick borne encephalitis increases in Sweden. Together with an increased awareness of the possibility to acquire protection by vaccination, this has led to an increase in the number of doses of the vaccine distributed in Sweden each year - now being approximately 400.000. The first year, two doses with an interval of 1 month is recommended for the general population, followed by a third dose approximately one year later and an additional booster dose three years after the third.

Preliminary results from a previous study showed a higher percentage protected (=titer at least 10) after 3 doses than after 2 doses (Rombo et al. EUDRA CT 2011 001348-31, unpublished information). In the same study, there were no differences between those who were vaccinated 0+7+21 compared to 0+30+90. The investigators were surprised to find marked differences between 2 and 3 doses also in the younger control group.

The investigators therefore aim to confirm results in a new study and to add a group with a double dose at day 0 and then a single dose at day 30 and 360

DETAILED DESCRIPTION:
The risk for tick borne encephalitis increases in Sweden. Together with an increased awareness of the possibility to acquire protection by vaccination, this has led to an increase in the number of doses of the vaccine distributed in Sweden each year - now being approximately 400.000. The first year, two doses with an interval of 1 month is recommended for the general population, followed by a third dose approximately one year later and an additional booster dose three years after the third.

The manufacturer of Encepur recommended a total of three doses to this age group using the same regimen as with "accelerated vaccination schedule (0+7+21 days). Unfortunately, geometrical mean of titers after 3 doses with the accelerated schedule is not superior to 2 doses given at 0+30 days The manufacturer of FSME-immune instead recommended that serology should be checked one month after the second dose and that a third dose should be given if titers are not sufficient (0+30+60 days). Unfortunately, determinations of titers in a large number of samples put severe strain on logistics and is not feasible in Sweden.

In order to try to improve immunity in the age group 60+ , the Department of Communicable Disease Control and Prevention in Stockholm therefore recommends a third dose two months after the first two doses to the age group 60+ (= 0+30+90 days).

Preliminary results from a previous study showed a higher percentage protected (=titer at least 10) after 3 doses than after 2 doses (Rombo et al. EUDRA CT 2011 001348-31, unpublished information). In the same study, there were no differences between those who were vaccinated 0+7+21 compared to 0+30+90. The investigators were surprised to find marked differences between 2 and 3 doses also in the younger control group

Primary aim: To study whether any differences remain before and one month after an additional dose at the following season Secondary aim: To study whether an additional dose of TBE vaccine 2 months after the second dose will improve protection in an age group 50+.

Primary endpoint: Serum concentration of neutralising antibodies against tick borne encephalitis one month after an additional dose the following year

Secondary endpoints: Serum concentration of neutralising antibodies against tick borne encephalitis one month after two or three doses.

Calculation of power: Depend on whether the aim is to determine differences in geometric mean titers or differences in seroconversion rate. The investigators prefer the former but have not settled for the least difference which would be interesting.

Inclusion critera: Age 50 years or more. Exclusion critera: previous tick borne encephalitis infection. Previously immunized with tick borne encephalitis vaccine. Anaphylactic reac tion to egg protein. Any disease or therapy which might suppress the immune response. Vaccination should be delayed if a participant has fever.

Study design. The investigators intend to give FSME-immune to 4 groups with varying vaccination schedules (see below) 50 participants will be randomized to each Group. A younger age group (50 participants between 18-49 years) will serve as controls and will be given FSME-immune according to standard recommendations (0+30 days)

Days 0 7 21 30 90 360 Vaccine group 1 x x x Vaccine group 2 x x x x Vaccine group 3 x x x x Vaccine group 4 xx x x Controls x x x

Blood samples (10 ml of blood) will be obtained for humoral response as shown below

Days 0 60 120 360 400 Group 1 x x x x x Group 2 x x x x x Group 3 x x x x x Group 4 x x x x x Controls x x x x x

Analyses Samples are analysed for neutralising antibodies at the Swedish institute for Infectious disease control - other options possible.

ELIGIBILITY:
Inclusion Criteria:

* Age 50 years or more (Control group 18 years)
* generally healthy
* no immunosuppressive condition
* fertile women must use contraceptives

Exclusion Criteria:

* Previous TBE infection
* Previously immunized with TBE vaccine
* Anaphylactic reaction to egg protein
* Any disease or therapy which might suppress the immune response
* Vaccination should be delayed if a participant has fever

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2015-01; Primary Completion 2016-02 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Serum concentration of neutralising antibodies against TBE one month after two or three doses. | 18 months after the first dose
  Determination of neutralising antibodies one month after completion of the first years vaccination series

SECONDARY OUTCOMES:
Serum concentration of neutralising antibodies against TBE one month after the dose which will be given a year later | 18 months after the first dose has been given
  Determination of neutralising antibodies one month after the dose which will be given a year later

CONTACTS AND LOCATIONS:
Overall Officials: lars rombo, MD, Principal Investigator — Karolinska Institutet
Locations (2):
- Dept infectious diseases, Helsinki, Finland
- Dept infectious diseases, Eskilstuna, Sweden